CLINICAL TRIAL: NCT01834963
Title: Randomised Phase II Study of Postoperative Hepatic Arterial Infusion Chemotherapy (Interferon/Fluorouracil Versus Low-dose Cisplatin/Fluorouracil) for Hepatocellular Carcinoma With Portal Vein Tumor Thrombus.
Brief Title: P2 Study of Postoperative Interferon/Fluorouracil vs Cisplatin/Fluorouracil for Hepatocellular Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHBO1207; UMIN000010425 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2017-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Interferon-alpha; Fluorouracil; CF regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interferon Alfa、Fluorouracil (Experimental): Interferon Alfa 5×10⁶International Unit(IU)/body subcutaneously 3 times a week for 4 weeks
  Fluorouracil 300mg/m2, day1-5,8-12, every 6 weeks
  Interventions: Drug: Interferon Alfa、Fluorouracil
- Cisplatin、Fluorouracil (Experimental): Cisplatin 20mg/m2 ,day1,8,22,29, every 6 weeks
  Fluorouracil 300mg/m2, day1-5,8-12,22-26,29-33, every 6 weeks
  Interventions: Drug: Cisplatin、Fluorouracil

INTERVENTIONS:
Drug: Interferon Alfa、Fluorouracil — Hepatic Arterial Infusion of 5-fluorouracil combined with systemic administration of Interferon-alpha
  Interferon Alfa 5×10⁶International Unit(IU)/body subcutaneously 3 times a week for 4 weeks
  Fluorouracil 300mg/m2, day1-5,8-12, every 6 weeks
  Other Names: Interferon Alfa ; IFN、; Fluorouracil ; 5-FU
  Arms: Interferon Alfa、Fluorouracil
Drug: Cisplatin、Fluorouracil — Hepatic Arterial Infusion of 5-fluorouracil and Cisplatin (Low-dose FP)
  Cisplatin 20mg/m2 ,day1,8,22,29, every 6 weeks
  Fluorouracil 300mg/m2, day1-5,8-12,22-26,29-33, every 6 weeks
  Other Names: Cisplatin ； Cispulan; Fluorouracil ; 5-FU
  Arms: Cisplatin、Fluorouracil

SUMMARY:
To evaluate the efficacy and safety of postoperative hepatic arterial infusion chemotherapy, interferon/fluorouracil versus low-dose cisplatin/fluorouracil, in patients with hepatocellular carcinoma with portal vein tumor thrombus.

DETAILED DESCRIPTION:
No standard treatment has been established for highly advanced hepatocellular carcinoma (HCC) invading the major branches of the portal vein except for sorafenib. Some reports suggested that hepatic arterial infusion chemotherapy improved survival of these patients. Other reports indicated surgical intervention improved that survival. However, there is no standard adjuvant therapy after liver resection for the patients with HCC with portal vein tumor thrombus in the main or first branch of the portal vein. Our preliminary results showed that combined interferon-alpha and intra-arterial 5-fluorouracil (5-FU) as a postoperative therapy prolonged disease-free and overall survival after liver resection. Hepatic arterial infusion chemotherapy using low-dose 5-FU and cisplatin is also promising regimen for advanced HCC.

Herein, the investigators planed the study to evaluate efficacy (two year survival as primary outcome, and overall-survival as secondary outcome) and safety ( as secondary outcome) in hepatic arterial infusion chemotherapy with continuous infusion of 5-fluorouracil and systemic administration of interferon-alpha or low-dose 5-FU and cisplatin, and to compare the efficacy as randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. hepatocellular carcinoma with histological or evidence or typical findings by CT or MRI.
2. surgically resectable tumors with tumor thrombus in first branch or main trunk of portal vein.
3. 20 years old or more.
4. Eastern Cooperative Oncology Group Performance status of 0 or 1.
5. Life expectancy of at least 6 months at the pre-treatment evaluation.
6. Child-Pugh class A or B.
7. Adequate bone marrow, liver and renal function, as assessed by the following laboratory requirements.

white blood cell count >= 2000/microliter, Neutrophil >= 1000/microliter, Hemoglobin >= 9.0 g/dL, Platelet count >= 75000/microliter, Total Bilirubin <= 1.5mg/dl, aspartate aminotransferase(AST) /alanine aminotransferase(ALT) <= 150 IU/L, Serum creatinine <= 1.2mg/dL, Creatinine clearance >= 60 ml/min

-

Exclusion Criteria:

1. Histological diagnosed combined hepatocellular and cholangiocellular carcinoma.
2. Extrahepatic tumor spread which affects patient's prognosis.
3. Hepatic encephalopathy
4. Active infections except for hepatitis B virus(HBV) and hepatitis C virus(HCV).
5. Sever complications (interstitial pneumonia, heart failure, renal failure, liver failure, ileus, incontrollable diabetes mellitus, and so on)
6. Active double cancer
7. Pregnancy 8-10) Medication or treatment that may affect to the absorption of drug or pharmacokinetics.

11) others, in the investigator's judgment.

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-02 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Two-year overall survival rate | Two years
  Duration: From randomization to evidenced death.
  Rate: Number of patients with evidenced death / number of total patients.
  2 year survival rate: survival rate at two-year from the randomization

SECONDARY OUTCOMES:
Progression free survival time | two years
  Progression free survival time from randomization to tumor progression based on RECIST or recurrence after curative surgery was calculated by Kaplan Meier methods.
Overall survival time | two years
  Overall survival time from randomization to evidence death was calculated by Kaplan Meier methods.
toxicity | At the end of hepatic arterial infusion chemotherapy (6 months)
  The incidence of adverse events evaluated by CTCAE Ver4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Nagano, MD, PhD, Study Director — Osaka University Graduate School of Medicine
Locations (1):
- Osaka University, Graduate School of Medicine, Osaka, Japan